CLINICAL TRIAL: NCT00267150
Title: Measurement of Patient Reported Gastrointestinal (GI) and Health-related Quality of Life (HRQL) Outcomes in Simultaneous Pancreas-Kidney Transplant Recipients
Brief Title: Gastrointestinal and Health-related Quality of Life Outcomes in Patients With Simultaneous Pancreas-Kidney Transplants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080ADE10
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Results first posted 2010-12-24 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Pancreas Transplantation; Kidney Transplantation
Keywords: Simultaneous Pancreas-Kidney Transplantation; mycophenolate; GI problems
MeSH Terms: interventions — Mycophenolic Acid

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Enteric-coated mycophenolate sodium (EC-MPS)

INTERVENTIONS:
Drug: Enteric-coated mycophenolate sodium (EC-MPS) — Experimental
  Other Names: myfortic

SUMMARY:
Treatment with the immunosuppressive drug mycophenolate mofetil (MMF) may result in gastrointestinal (GI) complications in some patients. This study will assess if a switch from MMF to enteric-coated mycophenolate sodium (EC-MPS) results in improved GI and/or health-related quality of life outcomes and determine the proportion of pancreas-kidney transplant recipients who experience any GI complaints under MMF-based immunosuppressive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Received simultaneous pancreas-kidney (SPK) transplant at least 3 months prior to study enrollment
* Receiving immunosuppressive regimen that includes MMF in combination with other immunosuppressive drugs (i.e., a calcineurin inhibitor, a mTOR inhibitor, steroids at least for three months at time of study enrollment)
* Receiving MMF for at least 1 month prior to enrollment; maximal MMF dose 2000 mg/d.

Exclusion Criteria:

* Patients with any known hypersensitivity to mycophenolic acid, mycophenolate sodium, mycophenolate mofetil or other components of the formulations (e.g. lactose; see also SCP of EC-MPS)
* If applicable, GI symptoms assumed or known to be induced by other drugs or infections (e.g. oral biphosphonates induced, infectious diarrhea)
* Acute rejection < 1 month prior to study enrollment

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2005-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Universitätsklinikum Charité Campus Virchow Klinikum Berlin Nephrologie und Internistische Intensivmedizin, Berlin, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Enteric Coated Mycophenolate-sodium: Enteric coated tablets of mycophenolate-sodium taken orally twice a day for 6-8 weeks.
Period: Overall Study
Arm/Group | Enteric Coated Mycophenolate-sodium
Started | 31
Completed | 30
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Enteric Coated Mycophenolate-sodium
Number analyzed (Participants) | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 48.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Changes in Gastrointestinal Symptom Severity and/or Health-related Quality of Life After Conversion From MMF to Enteric Coated Mycophenolate Sodium
Description: The Gastrointestinal symptom rating scale (GSRS) is a 15-item instrument designed to assess the symptoms associated with common gastrointestinal disorders. The GSRS has 5 subscales (reflux, diarrhea, constipation,abdominal pain, and indigestion) producing a mean subscale score ranging from 1 (no discomfort) to 7 (very severe discomfort). The GSRS total score was computed by the mean of the subscale scores. The primary analysis examined changes from Visit 1 (baseline) to Visit 2 (6-8 weeks) by computing the difference of GSRS total score.
Time Frame: weeks 6-8
Measure: Mean (Standard Deviation); unit: Change in Score of GSRS
Arm/Group | Enteric Coated Mycophenolate-sodium
Number analyzed (Participants) | 30
Change in Score of GSRS | -0.46 (0.71)

2. Secondary Outcome: Gastrointestinal Symptoms Under MMF-based Immunosuppressive Therapy
Description: Assessed by GI complications at baseline.
Time Frame: week 0
Population: Baseline population
Measure: Number; unit: Participants
Arm/Group | Enteric Coated Mycophenolate-sodium
Number analyzed (Participants) | 31
Participants
  Any complication | 19
  Diarrhea | 12
  Dyspepsia | 4
  Nausea | 3
  Abdominal pain/bloating/fullness | 11
  Other | 1

ADVERSE EVENTS:
Groups:
- All Patients: All patients
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 2/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=31)
Constipation (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.